CLINICAL TRIAL: NCT02859142
Title: Varenicline Augmentation of Patch Outcomes in Heavy Drinkers' Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-1615
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Results first posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Smoking Cessation; Alcohol Drinking
Keywords: Varenicline
MeSH Terms: conditions — Smoking Cessation; Alcohol Drinking | interventions — Varenicline; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Augmented Treatment (Experimental): Participants receive 12 weeks of Chantix along with standard smoking cessation treatment of nicotine patches and behavioral counseling visits.
  * Chantix (Varenicline) and NicodermCQ (Nicotine Patches): Administered according to package insert directions
  * Behavioral Counseling Sessions: Participants will attend one-on-one behavioral counseling sessions with a trained therapist at each of 4 study visits (pre-quit, quit date, week 2, and week 12). Behavioral sessions will involve teaching behavioral skills to assist with smoking cessation, preventing relapse, and coping with physical or emotional changes associated with cravings.
  Interventions: Drug: Chantix; Behavioral: Behavioral Counseling Sessions; Drug: NicodermCQ
- Standard Treatment w/ placebo (Active Comparator): Participants receive 12 weeks of standard smoking cessation treatment of nicotine patches and behavioral counseling visits in addition to placebo pills identical in appearance to varenicline
  * Placebo pills (identical to varenicline)
  * NicodermCQ (Nicotine Patches): Administered according to package insert directions
  * Behavioral Counseling Sessions: Participants will attend one-on-one behavioral counseling sessions with a trained therapist at each of 4 study visits (pre-quit, quit date, week 2, and week 12). Behavioral sessions will involve teaching behavioral skills to assist with smoking cessation, preventing relapse, and coping with physical or emotional changes associated with cravings.
  Interventions: Behavioral: Behavioral Counseling Sessions; Drug: NicodermCQ; Drug: Placebo

INTERVENTIONS:
Drug: Chantix — Chantix given alongside standard smoking cessation treatment, and administered per manufacturer's instructions [0.5 mg once per day for Days 1 to 3, 0.5 mg twice per day for Days 4 to 7, then one 1.0 mg tablet twice per day]
  Other Names: Varenicline Tartrate
  Arms: Augmented Treatment
Behavioral: Behavioral Counseling Sessions — One-to-one behavioral counseling sessions with a trained therapist
Drug: NicodermCQ — Nicotine patches provided over 12 week participation
  Other Names: Transdermal Nicotine Patch
Drug: Placebo — Identical in appearance to varenicline [0.5 mg once per day for Days 1 to 3, 0.5 mg twice per day for Days 4 to 7, then one 1.0 mg tablet twice per day]
  Arms: Standard Treatment w/ placebo

SUMMARY:
The purpose of this study is to learn if the combination of a study drug and patch is more effective in helping heavy drinkers stop smoking than just the patch alone The study drug, varenicline, has been approved by the Food and Drug Administration (FDA) to help people stop smoking, but it is not known if the addition of varenicline to standard smoking cessation treatment with nicotine patches will help people stop smoking who are regular, frequent drinkers. This study is being done because cigarette smoking is the number one preventable cause of death and disease in the United States.

DETAILED DESCRIPTION:
This study will conduct a real-world clinic-based smoking cessation trial examining the augmentation strategy of Chantix (Varenicline Tartrate), nicotine patch, and behavioral counseling versus standard treatment of patch plus behavioral counseling only in heavy drinkers who smoke (HDS). While Chantix is approved for smoking cessation, it is not routinely given in practice for HDS patients

In this study, there will be 4 total in-person study visits over the trial (pre-quit, quit date, week 2 and week 12), ending 12 weeks after the quit date. Biochemical verification from breath tests for CO, as well as vital signs and weight, will be measured at each visit along with survey responses measuring smoking urge and withdrawal, negative affect, neurocognition, and alcohol and smoking behaviors. These will also be used at a 26-week follow-up by telephone with biochemical verification for CO in those reporting being smoke-free.

Screening and Randomization Participants will respond to advertisements and will undergo a brief phone screening to determine initial eligibility requirements. Qualified candidates will be invited into the lab to conduct a short screening and study information session at the Clinical Addictions Research Laboratory at the University of Chicago. At screening, participants will sign an informed consent document. Next, demographics, smoking, alcohol and substance use patterns, health history, medications, vital signs, a urine test (for pregnancy and/or drug toxicology) and a blood test will be obtained.

Eligible participants will be randomized into one of two treatment groups: Standard Treatment (w/ placebo) will proceed with the study receiving nicotine patches and brief counseling sessions; Augmented Treatment will proceed with the same nicotine patches and brief counseling sessions, but will also receive standard dosing of Chantix (Varenicline tartrate).

Nicotine Patches Nicotine patches will be utilized starting at study quit date, and proceed according to package insert directions (10+ cigs/day smokers will begin with 21mg patches for six weeks, followed by 14mg patches for four weeks, and finally 7mg patches for two weeks. Those smoking fewer than 10 cigarettes/day will follow the same process starting at the 14mg patch level.

Chantix (Varenicline Tartrate) Those receiving Augmented Treatment will receive varenicline. They will undergo an up-titration week prior to the quit date, 12 weeks of target dosing, and a down-titration week. As per Pfizer recommendations, up-titration will be 0.5mg tablets once daily for 3 days followed by twice daily for four days leading to the quit date on day 8. The sequence will reverse for a down-titration week on week 13.

Placebo for Varenicline Those receiving standard treatment will also receive placebo medication that will be identical in appearance to and follow the same distribution protocol as varenicline.

Smoking Cessation Behavioral Sessions:

Participants will attend one-on-one behavioral counseling sessions with a trained Masters or PhD. Level therapist at each study visit. Behavioral sessions will involve teaching behavioral skills to assist with smoking cessation, preventing relapse, and coping with physical or emotional changes associated with cravings. At each study visit, subjective measures (i.e. brief self-report surveys about

Follow-Up Interview (Week 26) At Study Week 26, participants will complete a follow-up telephone interview, completing similar subjective measures as those completed during study visits. Participants reporting being smoke-free during this interview will arrange for biochemical verification of this status via expired CO testing either by arranging for a time to stop into one of the study sites or by arranging for study staff to meet with them in their home or workplace.

ELIGIBILITY:
Inclusion Criteria:

* Smoke 3-30 cigarettes/day
* Desire to quit smoking as indicated on a smoking stages ladder
* Consume >14 (men) or >7 (women) standard alcohol drinks per week (e.g., 1 drink = 12 oz beer, 5 oz wine, 1.5 oz liquor)
* Ability to understand, read, and write in English, at least 8th grade education
* Willing and able to sign an informed consent
* Stable residence and contact information.

Exclusion Criteria:

* Hepatic panel indices > 2 SD
* History of seizures or DTs during alcohol withdrawal
* Unstable medical (e.g., hepatitis, cirrhosis, seizure disorder, recent major cardiovascular event, etc.) or psychiatric disorder (e.g., active hallucinations, severe depression, obsessional thinking, self-injury risking significant blood loss, etc.) deemed by the study physician to be at significant risk for adverse interactions with study medications or measures.
* History of adverse reactions to varenicline (VAR) or nicotine patch
* Current suicidal ideation (past 6 months) and/or history of major suicide attempts.
* For women of child-bearing potential: currently pregnant, lactating, current plans to become pregnant in next three months, or unable to agree to adequate birth control during study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea King, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- Clinical Addictions Research Laboratory, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coe JW, Brooks PR, Vetelino MG, Wirtz MC, Arnold EP, Huang J, Sands SB, Davis TI, Lebel LA, Fox CB, Shrikhande A, Heym JH, Schaeffer E, Rollema H, Lu Y, Mansbach RS, Chambers LK, Rovetti CC, Schulz DW, Tingley FD 3rd, O'Neill BT. Varenicline: an alpha4beta2 nicotinic receptor partial agonist for smoking cessation. J Med Chem. 2005 May 19;48(10):3474-7. doi: 10.1021/jm050069n. PMID 15887955
- [Background] Perkins KA, Mercincavage M, Fonte CA, Lerman C. Varenicline's effects on acute smoking behavior and reward and their association with subsequent abstinence. Psychopharmacology (Berl). 2010 May;210(1):45-51. doi: 10.1007/s00213-010-1816-9. Epub 2010 Mar 20. PMID 20306175
- [Background] Tapper AR, McKinney SL, Nashmi R, Schwarz J, Deshpande P, Labarca C, Whiteaker P, Marks MJ, Collins AC, Lester HA. Nicotine activation of alpha4* receptors: sufficient for reward, tolerance, and sensitization. Science. 2004 Nov 5;306(5698):1029-32. doi: 10.1126/science.1099420. PMID 15528443
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Koegelenberg CF, Noor F, Bateman ED, van Zyl-Smit RN, Bruning A, O'Brien JA, Smith C, Abdool-Gaffar MS, Emanuel S, Esterhuizen TM, Irusen EM. Efficacy of varenicline combined with nicotine replacement therapy vs varenicline alone for smoking cessation: a randomized clinical trial. JAMA. 2014 Jul;312(2):155-61. doi: 10.1001/jama.2014.7195. PMID 25005652
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] King A, Vena A, de Wit H, Grant JE, Cao D. Effect of Combination Treatment With Varenicline and Nicotine Patch on Smoking Cessation Among Smokers Who Drink Heavily: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e220951. doi: 10.1001/jamanetworkopen.2022.0951. PMID 35244704
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902

RESULTS

PARTICIPANT FLOW:
Groups:
- Augmented Treatment: Participants received 12 weeks of Chantix along with standard smoking cessation treatment of nicotine patches and behavioral counseling visits.
  Drug: Chantix (Varenicline) Administered according to FDA approved package insert directions
  Drug: NicodermCQ (Nicotine Patches) Administered according to FDA approved package insert directions for 10 weeks
  Behavioral: Counseling Sessions Participants attended one-on-one behavioral counseling sessions with a trained therapist at the first 2 study visits [pre-quit day (medication initiation date, study week -1) and quit day (study week 0)]. Behavioral sessions involved teaching behavioral skills to assist with smoking cessation, preventing relapse, and coping with physical or emotional changes associated with cravings.
- Standard Treatment: Participants received 12 weeks of Placebo along with standard smoking cessation treatment of nicotine patches and behavioral counseling visits.
  Drug: Placebo (identical to Varenicline)
  Drug: NicodermCQ (Nicotine Patches) Administered according to FDA approved package insert directions for 10 weeks
  Behavioral: Counseling Sessions Participants attended one-on-one behavioral counseling sessions with a trained therapist at the first 2 study visits [pre-quit day (medication initiation date, study week -1) and quit day (study week 0)]. Behavioral sessions involved teaching behavioral skills to assist with smoking cessation, preventing relapse, and coping with physical or emotional changes associated with cravings.
Period: Overall Study
Arm/Group | Augmented Treatment | Standard Treatment
Started | 61 | 61
Completed (Completed indicates the number of participants completing the study, including those who discontinued medication but opted to remain in the study.) | 57 | 52
Not Completed | 4 | 9
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Scheduling difficulties | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Augmented Treatment: 12 weeks of active varenicline + 10 weeks of nicotine patches + behavioral counseling
  Chantix (Varenicline): Administered according to FDA approved package insert directions
  NicodermCQ (Nicotine Patches): Administered according to FDA approved package insert directions
  Behavioral: Counseling Sessions with a trained therapist at the first 2 study visits [pre-quit day (medication initiation date, study week -1) and quit day (study week 0)].
- Standard Treatment: 12 weeks of placebo + 10 weeks of nicotine patches + behavioral counseling
  Placebo (identical to Varenicline)
  NicodermCQ (Nicotine Patches): Administered according to FDA approved package insert directions
  Behavioral: Counseling Sessions with a trained therapist at the first 2 study visits [pre-quit day (medication initiation date, study week -1) and quit day (study week 0)].
- Total: Total of all reporting groups
Arm/Group | Augmented Treatment | Standard Treatment | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (12.89) | 44.02 (12.04) | 44 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 35 | 32 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 55 | 59 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 30 | 54
  White | 28 | 28 | 56
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 61 | 122
Duration of smoking in years [Mean (Standard Deviation); unit: years] | 25.5 (13.90) | 24.9 (12.62) | 25.2 (13.22)
Smoking days past month [Mean (Standard Deviation); unit: days] — Timeline Followback (TLFB) is a calendar-assisted interview in which participants report the number of cigarettes they consumed over a specified assessment period. Smoking Days is the total number of days participants reported smoking a cigarette during the 28 days prior to the screening visit.
  days | 27.84 (0.82) | 27.41 (1.68) | 27.6 (1.33)
Cigarettes per smoking day [Mean (Standard Deviation); unit: cigarettes] — Timeline Followback (TLFB) is a calendar-assisted interview in which participants report the number of cigarettes they consumed over a specified assessment period. Cigarettes per smoking day is the average number of cigarettes smoked per day on which any smoking was reported during the 28 days prior to the screening visit.
  cigarettes | 11.84 (6.26) | 11.66 (7.06) | 11.75 (6.65)
Fagerström Test for Cigarette Dependence score [Mean (Standard Deviation); unit: units on a scale] — Fagerstrom Test for Cigarette Dependence (FTCD) score is a standardized self-report measure used to assess for severity of cigarette smoking dependence. It consists of 6 items, with the two yes/no items scored from 0 to 1 and the four multiple-choice items scored from 0 to 3. A higher summary score (range: 0 - 10) indicates more severe cigarette dependence.
  units on a scale | 4.18 (2.36) | 3.64 (2.42) | 3.91 (2.40)
Expired carbon monoxide (CO) [Mean (Standard Deviation); unit: ppm] | 16.67 (11.32) | 17.54 (9.68) | 17.11 (10.50)
Alcohol drinking days [Mean (Standard Deviation); unit: days] — Timeline Followback (TLFB) is a calendar-assisted interview in which participants report how much alcohol they consumed over a specified assessment period. A trained interviewer records the number of standard drinks consumed on each day in the in the 28 days prior to the initial screening visit. Alcohol drinking days refers to the number of days on which any alcohol use occurred.
  days | 17.54 (7.07) | 18.90 (7.33) | 18.22 (7.20)
Drinks per drinking day past month [Mean (Standard Deviation); unit: drinks] — Timeline Followback (TLFB) is a calendar-assisted interview in which participants report how much alcohol they consumed over a specified assessment period. A trained interviewer records the number of standard drinks consumed on each day in the in the 28 days prior to the initial screening visit. Drinks per drinking day refers to the number of drinks consumed on days when any alcohol use occurred.
  drinks | 5.41 (3.73) | 6.08 (4.17) | 5.75 (3.95)
Heavy drinking days past month [Mean (Standard Deviation); unit: days] — Timeline Followback (TLFB) is a calendar-assisted interview in which participants report how much alcohol they consumed over a specified assessment period. A trained interviewer records the number of standard drinks consumed on each day in the in the 28 days prior to the initial screening visit. Heavy drinking was defined according to the National Institute on Alcohol Abuse and Alcoholism criteria of 5+ drinks for men and 4+ drinks for women.
  days | 8.28 (5.99) | 10.36 (8.77) | 9.32 (7.55)
DSM5 Alcohol use disorder severity [Count of Participants; unit: Participants] — Population: One participant from the Augmented Treatment group and one participant from the Standard Treatment group were missing DSM-5 AUD diagnosis data.
  Participants
    number analyzed (Participants) | 60 | 60 | 120
    None (0-1 symptoms) | 24 | 28 | 52
    Mild (2-3 symptoms) | 16 | 16 | 32
    Moderate (4-5 symptoms) | 14 | 9 | 23
    Severe (6+ symptoms) | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Smoking Abstinence Rates at 12 Weeks
Description: Number of participants reporting smoking abstinence at 12 weeks from baseline (smoking quit date) via subjective and biologically verified reports.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Augmented Treatment | Standard Treatment
Number analyzed (Participants) | 61 | 61
Participants | 27 | 17

2. Secondary Outcome: Change From Baseline in Self-Reported Alcohol Drinking Days at 12 Weeks
Description: Self-reported alcohol drinking days obtained via a past month Timeline Followback Calendar at 12 weeks
Time Frame: 12 weeks
Population: Study dropouts (i.e. lost to follow-up or voluntary withdrawals, N=13; 4 in augmented treatment and 9 in standard treatment groups) not include in means reported as drinking quantity and frequency are unknown.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Augmented Treatment | Standard Treatment
Number analyzed (Participants) | 57 | 52
days | 12.25 (9.54) | 11.96 (8.90)

3. Secondary Outcome: Change From Baseline in Self-Reported Alcohol Drinking Days at 26 Weeks
Description: Self reported monthly alcohol drinking days obtained via a past month Timeline Followback Calendar at 26 weeks
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Augmented Treatment | Standard Treatment
Number analyzed (Participants) | 57 | 52
days | 12.73 (9.06) | 11.44 (7.91)

4. Secondary Outcome: Change From Baseline in Self-Reported Heavy Drinking Days at 12 Weeks
Description: Self reported heavy drinking (5+ drinks/day for men, 4+ drinks/day for women) days obtained via a past month Timeline Followback Calendar at 12 weeks
Time Frame: 12 weeks
Population: Study dropouts (N=13; 4 in augmented treatment and 9 in standard treatment groups) not include in means reported as drinking quantity and frequency are unknown.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Augmented Treatment | Standard Treatment
Number analyzed (Participants) | 57 | 52
days | 5.02 (7.44) | 5.58 (7.54)

5. Secondary Outcome: Change From Baseline in Self-Reported Heavy Drinking Days at 26 Weeks
Description: Self reported heavy drinking (5+ drinks/day for men, 4+ drinks/day for women) days obtained via a past month Timeline Followback Calendar at 26 weeks
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Augmented Treatment | Standard Treatment
Number analyzed (Participants) | 57 | 52
days | 4.79 (5.33) | 5.56 (5.91)

6. Secondary Outcome: Change From Baseline Smoking Abstinence Rates at 26 Weeks
Description: Number of participants reporting smoking abstinence at 26 weeks from quit date via subjective and biologically verified reports.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Augmented Treatment | Standard Treatment
Number analyzed (Participants) | 61 | 61
Participants | 15 | 16

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each study visit (4 visits) over a 12 week period during active treatment.
Arm/Group | Augmented Treatment | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 2/61 | 0/61
Other Adverse Events (participants affected / at risk) | 59/61 | 48/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Augmented Treatment (N=61) | Standard Treatment (N=61)
Self-injurious thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Augmented Treatment (N=61) | Standard Treatment (N=61)
Nausea (Gastrointestinal disorders) | 34 | 18
Vomiting (Gastrointestinal disorders) | 9 | 3
Gas/flatulence (Gastrointestinal disorders) | 30 | 17
Abnormal dreams (Psychiatric disorders) | 45 | 30
Sleep problems (Psychiatric disorders) | 31 | 15
Increased heart rate (Cardiac disorders) | 10 | 6
Increased effects of alcohol (Psychiatric disorders) | 17 | 12
Suicidal thoughts (Psychiatric disorders) | 2 | 1
Dizziness (Nervous system disorders) | 12 | 12
Headache (Nervous system disorders) | 26 | 14
Joint pain (Musculoskeletal and connective tissue disorders) | 12 | 14
Skin irritation (Skin and subcutaneous tissue disorders) | 12 | 9
Other (General disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT02859142/Prot_SAP_000.pdf